CLINICAL TRIAL: NCT00346749
Title: A Randomized, Double-Blind, Parallel-Group, 12-Week Study to Evaluate the Anti-Inflammatory Effect of Fluticasone Propionate/Salmeterol DISKUS 250/50mcg BID Compared With Salmeterol DISKUS 50mcg Twice Daily in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: ADVAIR DISKUS® (Fluticasone Propionate/Salmeterol) Inhaler Versus SEREVENT DISKUS® (Salmeterol) Inhlaer On Inflammatory Cells And Markers In Chronic Obstructive Pulmonary Disease. ADVAIR DISKUS® and SEREVENT DISKUS® Inhalers Are Trademarks of the GSK Group of Companies.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated due to difficulties with finding sites and subjects willing to participate.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADC105931
Record Dates: First submitted 2006-06-28; First posted 2006-06-30 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Inflammation; FEV1; Sputum
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inflammation | interventions — Salmeterol Xinafoate; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Salmeterol; Drug: Fluticasone Propionate/Salmeterol Combination Product

INTERVENTIONS:
Drug: Salmeterol
Drug: Fluticasone Propionate/Salmeterol Combination Product
  Other Names: Salmeterol

SUMMARY:
This study evaluates the effect of two medicines on COPD (Chronic Obstructive Pulmonary Disease). The study will last 12 weeks. At the end of 12 weeks of treatment, subjects will stop the study medicines for 2 weeks. The study will involve 6 visits to the clinic. Subjects who elect to undergo bronchoalveolar lavage (BAL) procedures will have 8 study visits. Subjects will give sputum, blood, and in some cases BAL samples. Subjects will have breathing tests and will complete diary cards during the study. All study medicines and examinations will be given at no cost to the study subjects. Both medicines used in this study have been approved by the US FDA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD.
* Pre-bronchodilator FEV1 less than or equal to 70.0% and greater than or equal to 0.70L
* Ex-Smokers with at least a 10 pack-year history.

Exclusion Criteria:

* Current of secondary diagnosis of asthma or current diagnosis of atopy.
* Other respiratory disorders other than COPD.
* Other inflammatory diseases.
* Abnormal and clinically significant chest x-ray or ECG.
* Lung resection surgery within past 1 year.
* History of cancer not in remission within past 2 years.
* Serious, uncontrolled disease.
* Pregnancy or planning to become pregnant during the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2006-12; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Percent of sputum neutrophils

SECONDARY OUTCOMES:
Inflammation endpoints: Cell counts in sputum, cell counts and protein markers in BAL, protein markers in blood Clinical endpoints: FEV1 Airway conductance and airway resistance Functional residual capacity Shortness of breath symptoms

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- United States (10):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Fort Collins, Colorado
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: ADC105931 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: ADC105931 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: ADC105931 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: ADC105931 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: ADC105931 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: ADC105931 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register